CLINICAL TRIAL: NCT06204614
Title: Pilot Study of an Implantable Microdevice for in Situ Evaluation of Drug Response in Primary Bladder Tumors
Brief Title: Drug Screening Using IMD in Bladder Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Oliver Jonas, Director, Laboratory for Bio-Micro-Devices, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-269
Record Dates: First submitted 2023-12-11; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma
MeSH Terms: interventions — Methotrexate; Carboplatin; avelumab; Paclitaxel; Vinblastine; Gemcitabine; Cisplatin; Nivolumab; pembrolizumab; erdafitinib; enfortumab vedotin; sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- DRUG SCREENING USING IMD IN BLADDER CANCER (Experimental): Study participants placed in arm 1 will be implanted with the microdevice.
  Interventions: Device: Implantable Micro-Device; Drug: Methotrexate; Drug: Carboplatin; Drug: Avelumab; Drug: Paclitaxel; Drug: Vinblastine; Drug: Gemcitabine/Cisplatin I; Drug: Methotrexate/Vinblastine/Doxorubicin/Cisplatin/Avelumab; Drug: Gemcitabine/Cisplatin II; Drug: Cisplatin; Drug: Nivolumab; Drug: Pembrolizumab; Drug: Gemcitabine/Carboplatin; Drug: Methotrexate/Vinblastine/Doxorubicin/Cisplatin; Drug: Gemcitabine/Cisplatin/Nivolumab; Drug: Erdafitinib; Drug: Paclitaxel/Docetaxel/Ifosfamide; Drug: Gemcitabine; Drug: Gemcitabine/Carboplatin/Nivolumab; Drug: Enfortumab; Drug: Sacituzumab

INTERVENTIONS:
Device: Implantable Micro-Device — The implantable microdevice will release microdoses of specific drugs or drug combinations as a possible tool to evaluate the effectiveness of several cancer drugs against bladder cancer.
Drug: Methotrexate — Methotrexate will be placed in reservoir 1 of the implantable microdevice.
Drug: Carboplatin — Carboplatin will be placed in reservoir 2 of the implantable microdevice.
Drug: Avelumab — Avelumab will be placed in reservoir 3 of the implantable microdevice.
Drug: Paclitaxel — Paclitaxel will be placed in reservoir 4 of the implantable microdevice.
Drug: Vinblastine — Vinblastine will be placed in reservoir 5 of the implantable microdevice.
Drug: Gemcitabine/Cisplatin I — Gemcitabine/Cisplatin will be placed in reservoir 6 of the implantable microdevice.
Drug: Methotrexate/Vinblastine/Doxorubicin/Cisplatin/Avelumab — (Methotrexate/Vinblastine/Doxorubicin/Cisplatin/Avelumab) will be placed in reservoir 7 of the implantable microdevice.
Drug: Gemcitabine/Cisplatin II — Gemcitabine/Cisplatin will be placed in reservoir 8 of the implantable microdevice.
Drug: Cisplatin — Cisplatin will be placed in reservoir 9 of the implantable microdevice.
Drug: Nivolumab — Nivolumab will be placed in reservoir 10 of the implantable microdevice.
Drug: Pembrolizumab — Pembrolizumab will be placed in reservoir 11 of the implantable microdevice.
Drug: Gemcitabine/Carboplatin — Gemcitabine/Carboplatin will be placed in reservoir 12 of the implantable microdevice.
Drug: Methotrexate/Vinblastine/Doxorubicin/Cisplatin — (Methotrexate/Vinblastine/Doxorubicin/Cisplatin) will be placed in reservoir 13 of the implantable microdevice.
Drug: Gemcitabine/Cisplatin/Nivolumab — (Gemcitabine/Cisplatin/Nivolumab) will be placed in reservoir 14 of the implantable microdevice.
Drug: Erdafitinib — Erdafitinib will be placed in reservoir 15 of the implantable microdevice.
Drug: Paclitaxel/Docetaxel/Ifosfamide — (Paclitaxel/Docetaxel/Ifosfamide) will be placed in reservoir 16 of the implantable microdevice.
Drug: Gemcitabine — Gemcitabine will be placed in reservoir 17 of the implantable microdevice.
Drug: Gemcitabine/Carboplatin/Nivolumab — (Gemcitabine/Carboplatin/Nivolumab) will be placed in reservoir 18 of the implantable microdevice.
Drug: Enfortumab — Enfortumab will be placed in reservoir 19 of the implantable microdevice.
Drug: Sacituzumab — Sacitzumab will be placed in reservoir 20 of the implantable microdevice.

SUMMARY:
This research study involves implanting up to 4 microdevices, each small enough to fit inside the tip of a needle, into a tumor. These devices will release microdoses (many thousands of times less than a treatment dose) of different cancer drugs into the tumor. After approximately 72 hours, the devices and small regions of surrounding tissue will be removed and studied. There will be a follow-up visit within 42 days of device removal to assess for potential safety issues or side effects.

DETAILED DESCRIPTION:
This is a phase I pilot study of microdevice implantation and retrieval in patients with primary bladder cancer. The microdevice is 5x1mm and can be deployed using a biopsy needle placed percutaneously using imaging guidance. The purpose of the microdevice is to measure local intratumor response to antitumor medications in patients with primary bladder cancer. The microdevice contains multiple, separate reservoirs that are each loaded with a specific drug or drug combination.

Candidate patients will first be evaluated based on a CT or MRI, obtained as part of clinical care, and a physician who will determine whether the target lesion is amenable for microdevice implantation. Microdevice implantation will occur via cystoscopy using a flexible grasper (similar to that used for ureteral stent removal). Several independent microdevices will be placed per patient and target lesion. After implantation, the reservoirs release microdoses of each drug allowing the drug to interact with the tumor tissue in its native microenvironment. After device removal and before pathologic analysis, a repeat plain film X-ray of the bladder will be obtained to evaluate for microdevice migration. The microdevice(s) will be removed along with the target tumor as part of standard-of-care surgical excision. The tumor tissue surrounding the device will undergo pathologic and molecular analysis to assess local drug efficacy for each reservoir. These analyses will explore the impact of drug treatment on local cellular processes (e.g., apoptosis, pathway signaling).

The investigators will also investigate preliminary correlations between drug response as assessed by the microdevice and clinical outcomes and response to therapy. Collectively, these studies will establish the feasibility of clinical application of a drug-sensitivity microdevice in bladder cancer and the capacity of such a device to predict systemic response to cancer therapeutics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and the willingness to sign a written informed consent document.
2. Participants must have confirmed clinically localized bladder cancer with histology of urothelial cell carcinoma or variant histology and radiographic imaging consistent with stage T2-T3 N0 disease. Patients must be planned for cystectomy as part of their clinical care. The lesion planned for excision must be at least 1cm in size.
3. Participants must be 18 years of age or older. Patients must have the ability to understand and the willingness to sign a written informed consent document.
4. Participants must have confirmed clinically localized bladder cancer with histology of urothelial cell carcinoma or variant histology and radiographic imaging consistent with stage T2-T3 N0 disease. Patients must be planned for cystectomy as part of their clinical care. The lesion planned for excision must be at least 1cm in size.
5. Participants must be 18 years of age or older. Patients must have the ability to understand and the willingness to sign a written informed consent document.
6. Participants must have confirmed clinically localized bladder cancer with histology of urothelial cell carcinoma or variant histology and radiographic imaging consistent with stage T2-T3 N0 disease. Patients must be planned for cystectomy as part of their clinical care. The lesion planned for excision must be at least 1cm in size.
7. Participants must be 18 years of age or older.
8. Participants must be evaluated by a medical oncologist who will determine the clinically appropriate treatment strategy based on clinical history and extent of disease.
9. Patients must be deemed medically stable to undergo both percutaneous procedures and standard-of-care surgical procedures.
10. Participants will undergo laboratory testing within 30 days prior to the procedure (or within 72 hours if there has been a change in the clinical status since the initial blood draw). Patients must have absolute neutrophil count ≥1,000/mcL, platelets ≥50,000/mcL, PT (INR) 1.5 and PTT<1.5x control.
11. Participants must have undergone CT or MRI that assesses the extent of disease and allows the research team to assess for study eligibility. This will have been done as part of the standard-of-care.
12. The participant's case must be reviewed by the treating physician to assess the following factors:

    * Patient is clinically stable to undergo microdevice implantation and surgical procedures
    * Patient has sufficient volume of disease to allow implantation of the microdevice
    * Patient has a lesion for which the microdevice is a) amenable to percutaneous placement, and b) amenable to removal at the time of surgery
13. Patients must be willing to undergo research-related genetic sequencing (somatic and germline) and data management, including the deposition of de-identified genetic sequencing data in NIH central data repositories.
14. Patients must be agree to remain abstinent or use contraceptive measures for the duration of the study period

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit the safety of a biopsy and/or surgery.
2. Uncorrectable bleeding or coagulation disorder known to cause increased risk with surgical or biopsy procedures (detailed below in section 5.1.2.1).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-14 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety of microdevice placement and removal based on assessment of adverse events | From the time of arrival to interventional radiology for microdevice placement up to 6 weeks.
  A device will be declared safe if and only if all implanted devices do not cause an adverse event as defined in section 5.4. The device will be declared safe if 2 or less unacceptable toxicities are observed. Safety will be monitored using a BOIN-based boundary estimated assuming a 10% event rate and a stopping probability of 0.70. The boundary will not take effect until the third patient is enrolled. The trial will be stopped for safety concerns if the investigators see at least 1 adverse event in the first nine patients, or 2 adverse events across all 18. The probability of seeing 2 or less unacceptable toxicity events is 71% if the true rate of toxicity is 10% and 94% if the true rate of toxicity is 5%. The safety estimate will be summarized as number, percentage and with a 95% binomial confidence interval
Feasibility of microdevice placement | 48 Hours
  A placement is defined as successful if the investigators can implant and extract at least one microdevice from a patient's tumor with readable tissue for pathology from at least three-quarters of the device reservoirs surrounded by at least 400um of surrounding tissue. The investigators will declare feasibility if the lower bound of the 95% binomial CI does not exceed 0.65, that is if the investigators have 2 or fewer failures. The number of patients with successful retrieval will be summarized as number, percentage and with a 95% CI. Based on prior studies, if device reservoirs are surrounded by at least 400um of tissue, this enables downstream multi-omic analysis.

SECONDARY OUTCOMES:
Local intratumor response | 48 Hours
  To measure the local intratumor response to clinically relevant drugs in bladder cancer using quantitative histopathologic assessment of tumor tissue.
  The investigators will analyze tumor sections for each drug treatment zone using a immunohistochemical stain for apoptosis (cleaved caspase 3) and report the result for each condition as a percentage of positively stained cells (vs. total number of cells) within a radius of 500 microns from the drug reservoir.
  A board-certified pathologist will review staining quality of the histopathological staining.
Exploration of additional potential biomarkers of drug response | 48 Hours
  To explore additional potential biomarkers of drug response. We will perform immunohistochemical staining for markers of proliferation (ki67) and cell death (Cleaved Parp) in the local tumor tissue adjacent to the microdevice. Results will be calculated as a percentage of positively stained cells in the 500 micron radius adjacent to each reservoir on the microdevice, and will be reported as a percentage of positively stained versus total cells in the region of interest.
  Descriptive statistics will be used to summarize the results for each biomarker across multiple devices and drugs.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided